1. Title: In what way do music-based caregiving influence pain, daily activity, neuropsychiatric symptoms, and medication in patients with dementia?

Protocol approved by the Regional Comittees for Medical Research Ethics South East Norway, REK South East at **25.06.2019** 

NCT-number NCT04229446

ID: 2018/2519

#### 2. Introduction

The main objective of this study is to evaluate the pain-relieving effect of a well-characterized

non-pharmacological treatment program, music-based caregiving (MBC), to patients in

nursing homes with dementia and pain. This intervention study will apply for one  $\mbox{PhD}$ 

candidate. Patients with dementia disease will be recruited from eight different nursing homes

in Trondheim and Oslo, and each ward will be cluster randomized into intervention — or

control wards. Then the health care personnel in the intervention wards will receive education

in MBC and perform the intervention during eight weeks. The hypothesis is that this non-

pharmacological intervention will reduce pain intensity and improve the activity of daily

living (ADL), quality of life (QOL) and general activity, as well as reduce other symptoms in  $\,$ 

nursing home patients with dementia and pain compared to baseline.

#### Background

Pain is common in the elderly, and the prevalence of pain increase with age, co-morbidities

and frailty 1,2. While the prevalence of pain in older adults in the general population is

estimated to range from 25%-50% 2-4, the prevalence of pain in patients living in nursing

homes and community care varies from 28% to 87% 5,6. Musculoskeletal pain disorders have

been estimated to affect as many as 80% of those above 65 years 7.8. Although almost one

fifth of the elderly have symptomatic osteoarthritis 9, most of the chronic pain disorders are of

unknown cause 10. Thus opioids are not the best treatment with unclear effect over time and

serious side effects (sedation, dizziness, falls, dysphoria, obstipation) in the elderly 11. This

knowledge is in contrast to the practice today. In Denmark, 41% of nursing home residents

and 28% of home-domiciled patients with dementia use opioids 12.

Previous studies demonstrate that more than 80% of patients in nursing homes in

Norway had dementia disease 13,14. Dementia is a syndrome due to disease of the brain,

usually of a chronic and progressive nature, in which there is disturbance of multiple higher

cortical functions, including memory, reasoning, orientation, comprehension, calculation,

learning capacity, language, and judgement 15. Dementia has different stages; mild, moderate

and sever dementia. In severe dementia (disease), most of the patients have lost verbal

language and are dependent on of nursing care 15. Patients with dementia also experience

many severe neuropsychiatric symptoms. Selb $\tilde{A}$  k et al 16 followed 931 nursing home patients

with dementia over time. Agitation, irritability, disinhibition, and apathy were the most

prevalent and persistent symptoms during the study period. Depression and anxiety became

less severe over time, whereas the agitation subsyndrome (agitation /aggression, disinhibition,

and irritability) and apathy increased in severity during the follow-up period.

Pain is under-reported in the elderly since the elderly or the health care personnel do

not report pain, and because of failure of regular and systematic pain assessment in the health

care system 17. Pain assessment is challenging in the elderly because of impaired vision and

hearing, memory, verbal and cognitive functions, and neuropsychiatric symptoms. If not

adequately treated, chronic pain can cause depression, agitation, and aggression in patients

with dementia 18. Given the language loss in the most advanced stage of dementia and

sometimes after stroke, a cause of dementia, valid and reliable methods for pain assessment in

nonverbal older adults are needed 19. MOBID-2, an observation based pain assessment tool,

will be used in patients with dementia in the present study.  ${\tt MOBID-2}$  is validated in nursing

homes patients with dementia in Norway 6,20.

Based on current knowledge, non-pharmacological interventions should be the first-

line treatment approach for pain in most cases for patients with dementia 18. Since

pharmacological treatment for chronic pain is often inadequate and the elderly are prone to

side-effects, more evidence about non-pharmacological treatments is needed, especially for

elderly with dementia. Many studies are conducted in this area today, but unstructured and

non-evidence based interventions are commonly used 21 Based on current knowledge, non-

pharmacological interventions should be the first-line treatment approach for pain in most

cases for patients with dementia 18. Since pharmacological treatment for chronic pain is often

inadequate and the elderly are prone to side-effects, more evidence about  ${\tt non-}$ 

pharmacological treatments is needed, especially for elderly with dementia. Many studies are

conducted in this area today, but unstructured and non-evidence based interventions are  $\,$ 

commonly used 21. One of the most common non-pharmacological approaches for treating

behavioral and psychological symptoms of dementia is therapeutic use of music 22(. Many of

the studies done have low methodological quality with small sample sizes 23, but there seems

to be some evidence (for) that non-pharmacological interventions like activity and music can

relieve pain 24, depression25 and increase QoL 23. However, more research is needed using  $\,$ 

controlled studies of high quality 23.

The most convincing evidence of effect when reviewing interventions addressing QOL,

discomfort and behavior and psychiatric symptoms in person with dementia comes from

functional analysis-based interventions 26. These rely on the nursing home staff to implement

a care system, be involved in staff-education, protocol or systematic care planning. Examples

of such interventions are the ABC dementia, Serial-trial intervention and (the) TIME 27-29.

These interventions prove to be powerful and important systems to structure care-work,

deliverance and education, however they are comprehensive systems to implements and not

designed to inform on one specific symptom like pain. That is also why there is a shortage of

functional analysis-based interventions targeting pain intensity specifically.

The literature suggests that music may also provide effects for pain intensity for

patients with dementia 30. However, so far the studies are small, underpowered or performed

with less robust methods 31. A review that investigated whether interactive or receptive

deliverance (i.e. listening to) of music are more effective to reduce agitation in persons with

dementia found evidence that receptive deliverance does reduce agitation compared to

ordinary care, while interactive deliverance of music does not 32. In a recent review on non-

pharmacological treatments for individuals with dementia, sensory interventions like music

were most effective to reduce agitation followed by interventions targeting pain specifically

33. The evidence might suggest that music reduces stress due to sensory effects and by activating reminiscing.

Dhysical activity and active training has been i

Physical activity and active training has been investigated in persons with dementia

and have been able to prevent falls, improve physical and mental function and also

neuropsychiatric symptoms 34. There is currently a dearth of studies to provide information on

what interventions have proved to benefit pain intensity, and also looking at effects by age,

gender, type and grade of dementia 21. The physiological and psychological effects of music

have been thoroughly researched in later years. Precise therapeutic use of music can aid

attention, regulate autonomic dysregulation and access latent functional mental resources 35.

Music-based caregiving (MBC) has been developed through a dialogue between

neuroscience and clinical research in dementia care since the early 1990s, inspired by the

work of Michael Thaut and Linda Gerdner 36,37. Thaut and Gerdnerâ $\in$ TMs work has demonstrated

the clinical potential and efficacy of neurologic music therapy and individualized music 38.

 $\ensuremath{\mathsf{MBC}}$  has (been) continually built on neuroscientific research in continuing dialogue with the

Center for Biomedical Research at Colorado State University, Berklee School of

Music/Harvard Medical School in Boston and the neuroscientific work of  $T\tilde{A}\P$ res Theorell and

associates at Karolinska Sjukhuset in Stockholm 39. The PhD project - Integrated music in

nursing homes, an approach to dementia care, developed song, music and dance into a  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

systematic approach to dementia care through the period 2000â€~2012 40.

MBC provides in-

depth training on how music, song and movement can be used in caregiving for people with dementia. The program has been developed on behalf of the Norwegian

Directorate of Health and is based on neurological music therapy with elements of music

therapy and music education, and added to KompetanselÃ,ft 2020.

# 2.1 Need description

 $\ddot{\text{\sc i}}$  ,  $\cdot$  Increased focus on pain and non-pharmacological pain management in a vulnerable group

of patients

 $\ddot{\text{I}}$ . The non-pharmacological intervention can reduce pain intensity and strengthen ADL,

QOL and activity, reduce pharmacological side effects and reduce symptoms in nursing

home patients with dementia and pain without side effects.

ï,· Reliving pain without side effects will also be valuable for the patient's family.

 $\ddot{\textbf{r}}, \cdot$  This study will increase the focus on pain and pain management for health care

professionals in nursing homes and the community. The training of the staff in the

intervention nursing homes will enhance their clinical skills.

I,  $\cdot$  This increased competence can strengthen the motivation for the staff in the care of the

patients with dementia, and may reduce the turnover of the staff. Hopefully it can also

stimulate their wish for knowledge update.

 $\ddot{\mathbf{r}}$ . The health professionals in the intervention group will receive education in a program

with music, song and dance with the intention to reduce pain, and strengthen ADL,  ${\tt QOL}$ 

and activity, reduce side effects and reduce symptoms in nursing home patients with

dementia and pain. If the intervention shows effect, the health care professionals in the

control nursing homes will retain and, hopefully use, the training after the study is ended.

 $\ddot{i}$ , The research group is multi-professional from different research groups in Norway. All of

the nurses, physicians, experts in epidemiology, music therapy, and user participants work  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

together. This collaboration will strengthen the research competence for the group and for  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

the different members.

## 3.Aims and objectives

The overarching aim of the present study is to extend knowledge about pain in patients with  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

dementia and to evaluate if an intervention with music-based caregiving (MBC) will reduce

pain intensity and improve activity and QoL in nursing home patients with dementia and pain.

The baseline descriptions of pain and pain management in patients with dementia disease in  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

the included nursing homes will be published as a part of another study.

The research questions in the present study are:

1. Will music based caregiving reduce pain and the need for analgesics in patients with  $\ensuremath{\mathsf{N}}$ 

dementia in nursing homes?

2. Will music-based caregiving impact on QoL, ADL function, and total daily physical  $\,$ 

function?

3. Will implementation of music-based caregiving impact on neuropsychiatric symptoms and psychopharmacological medication?

The primary aim is to give better and safer pain management to patients with pain and dementia in nursing homes.

Secondary aims are:

- to increase total daily activity, ADL function, QoL, and reduce neuropsychiatric symptoms, and
- to increase knowledge of pain in patients in nursing homes: the occurrence, intensity, location, treatment, diagnoses, and comorbidities.

## 4. Project methodology

#### 4.1. Design, method and analysis

This is a cluster-randomized controlled trial including patients with dementia and pain living at different wards at eight nursing homes.

1) Eight nursing homes will be selected to participate, four in Trondheim and four in Oslo.

established with randomly selected nursing homes.

2) Subsequently, all patients at the 8 nursing homes will be screened with respect to  $\,$ 

dementia and pain (see screening tools later). If patients have dementia and report pain

(â%¥3 on MOBID) they will be included in the study.

3) The included patients will then have a clinical examination of pain and pain management

by an expert physician (see below). Evaluation of the use of analgesics psychopharmacological medication will be performed. Inappropriate medication (both too

much and too little) will be corrected in collaboration with the nursing home doctor.

4) In addition to the clinical examination of pain, we will measure total daily physical

activity, ADL, QOL, and neuropsychiatric symptoms on all included patients (see below).

- 5) After the pre test a randomization of the wards into intervention wards or control wards will be performed.
- 6) About 5 staff members at each of the wards randomized to the intervention group will

receive education in the MBC before intervention (see below).

7) As a post-test three month after the intervention has ended, pain, total daily physical

activity, ADL, QOL, and neuropsychiatric symptoms will be measured.

This design facilitates the measurement of the outcome variables in nursing homes patients

before and after the intervention, and between the two groups. The results from the pre- and  $\,$ 

post-tests will be compared between the groups to assess whether or not the intervention has

effects on the outcome variables when adjusting for baseline levels (pretest). This approach

will allow us to evaluate whether changes in the outcome measure are caused by the  $\,$ 

intervention or other elements.

## Participants

In total, 240 patients with dementia and pain (120 from nursing homes in Trondheim and 120

from nursing homes in Oslo) will participate in the study. Contact is already established with

nursing homes that will participate both places. Patients will be included if they report

moderate pain or more ( $\hat{a}\%$ ¥3 on MOBID) and mild dementia or more ( $\hat{a}\%$ ¥1 on CDR). They will

not be included if they have lived in the nursing home less than four weeks, have short (less

than eight weeks) expected lifetime (judged by the nurses), and if they do not understand the  $\$ 

Norwegian language. Anonymous data will be collected for comparing patients not included

with those included, and the reasons for why they were not included will be described. Before

inclusion in the study, patients or their relatives should give an informed consent.

#### Clinical examination

All the included patients will be clinically examined by expert physicians in the same way as

performed in the HUNT3 study 10. Focal pain conditions will be diagnosed according to the

 $10 \, \mathrm{th}$  revision of the International Statistical Classification of Diseases and Related Health

Problems 41, either as a disease diagnosis, or, if no cause of the pain can be identified, by a

pain/symptom diagnosis. In addition, the physician will make a critical evaluation of their

analgesic and other medications as mentioned above. If medications are inadequate, obviously

give side effects, or are in violation with current guidelines, the recommendation for

correction will be given to the physician at the nursing home. This procedure will particularly

be the case for all patients having a pain state of known origin with documented effect of

specific medication (i.e. osteoarthritis or neuropathic pain).

## Education of the health care professionals

After pre-test including clinical examination, a randomization of the wards into intervention

wards or control wards will be performed. About 5 staff members at each of the wards

randomized to the intervention group will receive education in the MBC. Approximately  $60\,$ 

employees will receive training in MBC by Myskja and  $H\tilde{A}$ pnes with a 5-day training course.

This training will facilitate the intervention in the way that the health professionals in the  $\$ 

intervention group will be competent in applying active (song, dance) and passive (music

listening) modalities in individualized music with groups and individuals as needed, mindful

of personal preference and dignity and aware of the sensory environment.

#### The MBC program

The MBC program has been developed as a hermeneutic circle (interpreted from the Vedic

scriptures) 42, expanding from literature reviews and teaching sites to observations of clinical

response, aided by video analyses. The Medical Research Council guidelines have been

followed in this process, using the cyclical stages of development, feasibility and piloting,

evaluation, and implementation 43. In the period from 2012, 490 health care workers have

been educated in this program in Trà ndelag.

#### Intervention

The intervention will be applied by the trained staff with daily individualized prerecorded  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

music integrated with activity with about 30 minutes duration, combined with a one hour

active session in groups twice weekly. The control group will receive regular treatment with

the same improved analgesic treatment as the intervention group, but without MBC. The  $\,$ 

duration of the intervention and the control period will be eight weeks.

#### Measurements

As a part of the pre-test we will select data about the patients  $\hat{a} \in \mathbb{T}^m$  demographics, diagnoses and medication use from the medical chart.

## Stage of dementia disease

Clinical Dementia Rating Scale (CDR) is an assessment scale for the accurate clinical staging

of dementia in older subjects. The CDR includes  $\sin$  items assessing cognitive and functional

impairment. Based on an algorithm giving precedence to the item memory a CDR total score

is estimated. A score of 0, 0.5, 1, 2, 3 indicates no dementia, questionable dementia, mild,

moderate or severe dementia, respectively, and CDR score > 1, is cut-off score for dementia

disease. The scale has shown to be reliable and valid and is translated into Norwegian  $\,$ 

language 44.

#### Pain

MOBID-2 pain scale will be used for pain assessment in elderly people with dementia 20,45.

The assessment of inferred pain intensity is observed based on patient  $\hat{a} \in \mathbb{T}^m$  s pain behaviors during

standardized, guided movements of different body parts (Part 1). In addition,  ${\tt MOBID-2}$ 

includes an observation of pain behavior related to internal organs, head and skin registered  $\,$ 

on pain drawings and monitored over time (Part 2). MOBID-2 has shown to be sufficiently

reliable, valid and time-effective to assess pain in patients with severe dementia  $46\,.$  We will

use MOBID-2 for assessment of pain in all the patients with dementia.

Quality of life and aids of daily living

Quality of Life in Late-Stage Dementia (QUALID) measures QOL in patients with severe

dementia based on information and observations from nurses about the patient  $\hat{a} \in \mathbb{T}^m$  s emotions and

behavior. The scale has been validated in a Norwegian nursing home population, showing

satisfactory psychometric properties 47,48.

Dementia Quality of Life (DQoL). Because QUALID-scale is an observation scale, and there

is a lack of studies comparing self-reported and observations QoL in those with dementia, we

want to compare the observation estimate with self-report for patients with none, mild and

moderate dementia (DQoL). DQoL consists of five domains: self-esteem, positive affect/  $\,$ 

humor, feeling of belonging, and sense of aesthetics and negative affect. The instrument is

evaluated in those with mild and moderate dementia and is used in nursing homes in Norway 49.

Barthelâ $\in$ <sup>TM</sup>s Activities of Daily Living Index (ADL) is a screening instrument for patientsâ $\in$ <sup>TM</sup> daily

life functioning. This 10-point scale measures patients  $\hat{\mathbf{e}}^{\text{m}}$  degree of self-reliance with a total

score ranging from 0 to 20. Lower scores indicate greater dependence on nursing care 50.

The total daily physical activity using two 3-axis accelerometers (Axivity, UK) attached to the

skin on the right thigh and low back for 7 continuous days. By utilizing state-of-the-art

machine-learning techniques, we have developed a preliminary activity recognition model for

lying, sitting, standing, walking and other activities. This model is being used in the Nord-

 ${\tt Tr\tilde{A}}_{\tt i}{\tt ndelag}$  health study (HUNT4). Specifically, the model captures walking velocity and

transitions between postures and activities (e.g. sit-to-stand) and sleep quality/duration.

Neuropsychiatric symptoms and depression

The Neuropsychiatric Inventory (NPI-NH) measure 12 different psychiatric symptoms and

behavioural disturbances in nursing home residents: delusions, hallucinations, dysphoria,

anxiety, agitation/aggression, euphoria, disinhibition,

irritability/lability, apathy, aberrant

motor activity, sleep and night-time behaviour disorders, appetite and eating disorders. The

screening question is asked to determine if the behavioural change is present. If a screening

question is present, there will be sub-questions about frequency (score 1 to 4) and intensity

(score 1 to 3) for each behavior. Total score for each behavior is from 1 to 12. The scale has

been validated for patients in nursing homes in Norway 51.

Cornell scale for depression in dementia assesses signs and symptoms of major depression in

patients with dementia in an interview with the health care providers. The scale consists of 19

items in five domains based on observation of behaviour 52. Each question is scored on a two-

point scale: 0=absent; 1=mild or intermittent; 2=severe; n/a = unable to evaluate 2.

#### Sample size

A power calculation was performed on MOBID-2. Based on the literature review we assumed

the mean difference to be 1.2 and the common standard deviation to be 3. To keep statistical

power of 80% (beta = 0.2) and significance level of 5%, we would need 100 in each group to

reveal the anticipated difference between the groups as statistically significant. Taking in

consideration the possible cluster effect of 20% we aim to enrol 120 patients in both groups 20,53,54.

## Statistical analyses

Participants  $\hat{\mathbf{a}} \in \mathbb{M}$  background characteristics will be described as means and standard deviations

(SD) for normally distributed continuous data or medians and range for continuous data with

skewed distributions. Categorical data will be presented as counts and percentages. At the pre-

test, possible between-group differences will be assessed using independent samples t-tests

when comparing pair of normally distributed continuous variables, chisquare test for

categorical variables and Mannâ $\in$  "Whitney test for continuous variables with skewed

distribution. Possible differences between the groups concerning the mean  ${\tt MOBID-2\ Pain}$ 

Scale, QoL, ADL, total daily physical activity, and neuropsychiatric symptoms scores over

time and at given time points will be estimated with linear random intercept quantile mixed-

effect models. Mixed model regression modelled with linear random intercept permits

multiple measurements per person over time, irregular intervals between measurements and  $% \left( 1\right) =\left( 1\right) +\left( 1\right) +\left$ 

allows for incomplete data on assumption that data are missing at random 55. A significance

level of 5 % will be considered statistically significant for all analyses. Data will be analyzed

using IBM Statistical Package for the Social Sciences (SPSS) version 23.

## 4.2. Participants, organization and collaboration

The multi-professional research group will unite clinical and scientific experience from four

different universities (for more details and contribution to the study, see e-application):

Petter Chr. Borchgrevink, MD, PhD (principal investigator, main supervisor). Leader of "Pain

research group". Head of "Dept of Pain and Complex Disorders" at  $\mathrm{St.Olav}\hat{A}$ 's Hospital and

Professor of Anesthesiology and Pain Management at NTNU. Leader of the Norwegian  $\ensuremath{\mathsf{Dept}}$ 

of Health-defined "Pilot Project for Joint Multidisciplinary Diagnosis Centers / Outpatient

Clinics for Patients With Chronic Pain and/or Fatigue Disorders of unknown cause". Has 118

scientific publications and supervised 9 candidates on their PhD.

Tone Rust $\tilde{\text{A}}$  en Professor, RN, PhD (co supervisor). She has 128 scientific publications, and

has been the main supervisor for 12 PhD candidates that have completed their PhD. Rust  $\tilde{\text{A}}_{\text{s}}$  en

is a professor at University of Oslo and a researcher at Oslo University Hospital. She has a

long experience with pain research and is the leader of the Regional Research Network

NORSMAN funded by Helse SÃ, rà st.

Karin Torvik RN, PhD. Associate professor, NTNU, Nord University, Faculty of Health and

Nursing, Levanger, Norway (co-supervisor). She has a long experience in guiding master and  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

bachelor students. Her research area is pain assessment and pain management in the elderly.

Geir Selbæk MD, PhD, professor (co supervisor): He has 134 scientific publications. He has

supervised 7 candidates on their PhD, and is currently supervising 10 PhD candidates. He is

the primary investigator for several large-scale clinical studies, nationally and internationally.

His research experience spans a wide variety of fields including basic medicine,

epidemiological studies, clinical trials. This year he was awarded the Norwegian dementia

research prize by the Norwegian Health Association.

Audun Myskja MD, PhD. Advisor to The Norwegian National Resource Center for Arts and

Health. He is a strong and important voice in the traditional academic setting, seeking to

create simple practice-based methods to connect science and the fields of the common human

experience, expanding the context of traditional Western medicine. He has long experience

with innovative use of musical elements in rehabilitation of dementia and  $Parkinson \hat{a} \in \mathbb{T}^m s$ 

patients, and for creating systematic tools for empowerment in persons with chronic illness.

Vegar Rangul PhD, Associate professor/Post.doc. HUNT Research Centre, Department of

Public Health and Nursing, Faculty of Medicine, NTNU. Is a specialist in physical activity

epidemiology and has extensive experience with the use of large epidemiological data sets to

resolve issues relating the health effects of physical activity and their interaction with general

health behavior and cardiovascular disease risk in particular. Has expertise in behavioral  $% \left( 1\right) =\left( 1\right) +\left( 1\right)$ 

epidemiology, measurement of physical activity and epidemiological population studies.

Odd H $\tilde{\text{A}}$ ¥pnes, General manager of the Norwegian Resource Center for Arts and Health, NORD

University. He holds a master of musicology, education-in-science and education and has

been central in the development of MBC as a national program. He has been the head of the

national node for culture and health 2000-2003, and participates in international cooperation and research networks in Arts and Health.

Reidun Sandvik RN, PhD. Associated professor, Western Norway University of Applied

Sciences and University of Bergen. She has experience with supervising master students. Her

PhD topic was pain in nursing home patients with dementia and she has continued with

research about pain management for this group of patients.

Milada C  $Sm\tilde{A}Ystuen$  PhD, biostatistician. Will help with data management and statistical analyses for the whole study and all three papers.

# 4.3. Budget

We will apply for one doctoral student. For details se the electronic application (es $\tilde{A}_{\mbox{\tiny $\lambda$}}$ knad).

4.4. Plan for activities, visibility and dissemination

Timeline - see electronic application

Publication plan The most important results to emerge from the project will be disseminated through different channels. The PhD student will write 3 scientific papers:

- a) The effect of music based caregiving on pain and the need for analgesics in patients with dementia in nursing homes.
- b) The effect of music-based caregiving on QoL, ADL function, and total daily physical function.
- c) The effect of music-based caregiving on neuropsychiatric symptoms and psychopharmacological medication.

Workshop, seminars and conferences: It is important that leaders in community health care

and individuals in charge of nursing homes have access to our results. To facilitate this, we

will arrange workshops and seminars to present our results. The PhD student will participate

in at least two international and one national conference during their study period, presenting  $% \left( 1\right) =\left( 1\right) +\left( 1\right) +\left($ 

her/his work.  $\hat{a} \in \infty Nasjonal for eningen for folkehelsen <math>\hat{a} \in \infty Nasjonal for eningen for folkehelsen \hat{a} \in \infty Nasjonal for eningen for folkehelsen <math>\hat{a} \in \infty Nasjonal for eningen for folkehelsen \hat{a} \in \infty Nasjonal for eningen for eningen for folkehelsen \hat{a} \in \infty Nasjonal for eningen for e$ 

#### 4.5. Plan for implementation

As the study is an intervention study it can easily be implemented into practice if the results

are positive. The results from the present study will also be transferable to other patient

groups that cannot communicate their pain. The findings from the present study will be  $\frac{1}{2} \int_{\mathbb{R}^{n}} \frac{1}{2} \left( \frac{1}{2} \int_{\mathbb{R}^{n}} \frac{1}{2} \left( \frac{1}$ 

relevant outside nursing homes as these patients also are in specialist hospitals and in the community.

#### 5. User involvement

Hans  $H\tilde{A}_{,,j}$ gh Henrichsen is user participant from Oslo Municipal. He has been informed about

Municipality (Torunn Vatne). From Trondheim, one patient with dementia and one relative of

one patient with dementia will be recruited from the Resource Center for Dementia Disease in

Trondheim and will be user participants. All participants will be involved in the detail

planning of all phases of the project. The National Association for Public Health, which has

given feedback on the application, will also recruit user participants from the local dementia  $\frac{1}{2}$ 

associations if the study should be funded.

# 6. Ethics

After permission to include the nursing homes, meetings will be arranged with the staff to

inform and motivate them for carrying out the study. The health care providers will collect

written or oral informed consent from the patients and/or their legal guardians or relatives. We

will use different inclusion procedures depending on the patients  $\hat{a} \in \mbox{}^{\text{\tiny{TM}}}$  consent competence in

collaboration with the Ethical Committee.

Patients with consent competence will receive oral and written information prior to the study,

and the nurses will obtain written informed consent. If the patients cannot sign, they will give

oral consent to the nurse, and the nurse will sign the informed consent on behalf of the

patients. If the patients are cognitively impaired, guidelines from the Ministry of Health and

Care Service in Norway will be followed when recruiting these patients. Relatives of patients  ${\bf r}$ 

or their legal guardians will receive written information prior to the study and consent on their

behalf. The cognitively impaired patients will receive oral information prior to the study and

will not be included if they decline to participate, even if their relatives/legal guardians had consented on their behalf.

One can ask if it is unethical to not give music therapy to all included patients in the  $\$ 

nursing homes. However, we are not taking away anything from the patients, and all included participants will receive pain assessment.

#### 7. References

- 1.Cooper JW, Burfield AH. Assessment and management of chronic pain in the older adult. J Am Pharm Assoc (2003) 2010; 50(3): 89-99.
- 2.Rustã en T, Wahl A, Hanestad B, Lerdal A, Paul S, Miaskowski C. Age and the experience of chronic pain: differendes in health and quality of life among younger, middel-aged and older audults. Clin J Pain 2005; 21: 513-23.
- 3.American Geriatrics Society. The management of persistent pain in older persons. J Am Geriatr Soc 2000; 40: 205-24.
- 4. Johannes CB, Le KT, Zhou X, Johnston JA, Dworkin RH. The prevalence of chronic pain in United States audults: results of n internet based survey. J Pain 2010; 11(11).
- 5. Sandvik RK, Selbaek G, Seifert R, et al. Impact of a stepwise protocol for treating pain on pain intensity in nursing home patients with dementia: a cluster randomized trial. Eur J Pain 2014; 18(10): 1490-500.
- 6.Torvik K, Kaasa S, Kirkevold O, Rustoen T. Pain in patients living in Norwegian nursing homes. J Palliat Med2009;23:8-16.

- 7.Boeckxstaens P, Peersman W, Goubin G, et al. A practice-based analysis of combinations of diseases in patients aged 65 or older in primary care. BMC Fam Pract 2014; 15: 159.
- 8.Won A, Lapane K, Gambassi G, Bernabei R, et al. Correlates and management of nonmalignant pain in the nursing home. SAGE Study Group. Systematic Assessment of Geriatric drug use via Epidemiology. J Am Geriatr Soc 1999; 47(8): 936-42.
- 9. Jordan JM, Helmick CG, et al. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol 2007; 34: 172-80.
- 10.Glette M, Landmark T, Jensen MP, et al. Catastrophizing, Solicitous Responses From Significant Others and Function in Individuals with Neuropathic Pain, Osteoarthritis or Spinal Pain in the General Population. J Pain 2018.
- 11.Barber JB, Gibson SJ. Treatment of chronic non-malignant pain in the elderly: safety considerations. Drug Saf 2009; 32: 457-74.
- 12.Jensen-Dahm C, Gasse C, Astrup A, Mortensen PB, Waldemar G. Frequent use of opioids in patients with dementia and nursing home residents: A study of the entire elderly population of Denmark. Alzheimer's & dementia: the journal of the Alzheimer's Association 2015; 11(6): 691-9.
- 13.Bergh S, Holmen J, Saltvedt I, Tambs K, Selbæk G. Dementia and neuropsychiatric symptoms in nursing-home patients in Nord-TrÃ, ndelag County. Tidsskr Nor Laegeforen 2012; 132(17): 1956-9.
- 14.Helvik AS, K E, J.Š. B, Selbæk G. Prevalence and Severity of Dementia in Nursing Home Residents. Dement Geriatr Cogn Disord 2015; 40(3-4): 166-77.
- 15.Centers for disease control and prevention. International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM). 18.08.2017 2017. https://www.cdc.gov/nchs/icd/icd10cm.htm (accessed 16.05 2018).
- 16.Selbaek G, Engedal K, Benth JS, Bergh S. The course of neuropsychiatric symptoms in nursing-home patients with dementia over a 53-month follow-up period. Int Psychogeriatr 2014; 26(1): 81-91.
- 17. Miaskowski C. The impact of age on a patient's perception on pain and ways it can be managed. Pain Manag Nurs 2000; 1: 2-7.
- 18. Malara A, De Biase GA, Bettarini F, et al. Pain Assessment in Elderly with Behavioral and Psychological Symptoms of Dementia. J Alzheimers Dis 2016; 50(4): 1217-25.
- 19. Kaasalainen S. Pain assessment in older audults with dementia. Using behavioral observation methods in clinical practice.

- Careful use can guide decision making and improve care. J Geront Nurs 2007; 33(6): 6-10.
- 20. Husebo BS, Strand LI, Moe-Nilssen R, Husebo SB, Ljunggren AE. Pain in older persons with severe dementia. Psychometric properties of the Mobilization-Observation-Behaviour-

Intensity-Dementia (MOBID-2) Pain Scale in a clinical setting. Scand J Caring Sci 2010; 24(2): 380-91.

- 21.Garrido S, Dunne L, Chang E, Perz J, Stevens CJ, Haertsch M. The Use of Music Playlists for People with Dementia: A Critical Synthesis. J Alzheimers Dis 2017; 60(3): 1129-42.
- 22.Pedersen SKA, Andersen PN, Lugo RG, Andreassen M, Sutterlin S. Effects of Music on Agitation in Dementia: A Meta-Analysis. Front Psychol 2017; 8: 742.

- 23.Abraha I, Rimland JM, Trotta FM, et al. Systematic review of systematic reviews of non-pharmacological interventions to treat behavioural disturbances in older patients with dementia. The SENATOR-OnTop series. BMJ Open 2017; 7: e012759.
- 24. Park H. Effect of music on pain for home-dwelling persons with dementia. Pain Manag Nurs 2010; 11(3): 141-7.
- 25.Pongan E, Tillmann B, Leveque Y, et al. Can Musical or Painting Interventions Improve Chronic Pain, Mood, Quality of Life, and Cognition in Patients with Mild Alzheimer's Disease? Evidence from a Randomized Controlled Trial. J Alzheimer's disease 2017; 60(2): 663-77.
- 26. Dyer SM, Harrison SL, Laver K, Whitehead C, Crotty M. An overview of systematic reviews of pharmacological and non-pharmacological interventions for the treatment of behavioral and psychological symptoms of dementia. Int Psychogeriatr 2017: 1-15.
- 27.Rokstad AM, Rosvik J, Kirkevold O, Selbaek G, Saltyte Benth J, Engedal K. The effect of person-centred dementia care to prevent agitation and other neuropsychiatric symptoms and enhance quality of life in nursing home patients: a 10-month randomized controlled trial. Dement Geriatr Cogn Disord 2013; 36(5-6): 340-53.
- 28.Lichtwarck B, Selbaek G, Kirkevold O, et al. Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropsychiatric Symptoms: A Cluster Randomized Controlled Trial. Am J Geriatr Psychiatry 2017.
- 29.Kovach CR, Logan BR, Noonan PE, et al. Effects of the Serial Trial Intervention on discomfort and behavior of nursing home residents with dementia. Am J Alzheimers Dis Other Demen 2006; 21(3): 147-55.
- 30.Dyer SM, Harrison SL, Laver K, Whitehead C, Crotty M. An overview of systematic reviews of pharmacological and non-pharmacological interventions for the treatment of behavioral and psychological symptoms of dementia. Int Psychogeriatr 2018; 30(3): 295-309.
- 31. Pieper MJ, van Dalen-Kok AH, Francke AL, et al. Interventions targeting pain or behaviour in dementia: a systematic review. Ageing Res Rev 2013; 12(4): 1042-55.
- 32. Tsoi KKF, Chan JYC, Ng YM, Lee MMY, Kwok TCY, Wong SYS. Receptive Music Therapy Is More Effective than Interactive Music Therapy to Relieve Behavioral and Psychological Symptoms of Dementia: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc 2018.
- 33.Legere LE, McNeill S, Martin LS, Acorn M, An D. Non-pharmacological approaches for behavioural and psychological symptoms of dementia in older adults: A systematic review of reviews. J Clin Nurs 2017.

- 34. Hoffmann K, Sobol NA, Frederiksen KS, et al. Moderate-to-High Intensity Physical Exercise in Patients with Alzheimer's Disease: A Randomized Controlled Trial. J Alzheimers Dis. 2016; 50(2): 443-53.
- 35.Livingston G, Kelly L, Lewis-Holmes E, et al. Non-pharmacological interventions for agitation in dementia: systematic review of randomised controlled trials. Br J Psychiatry 2014; 205(6): 436-42.
- 36. Thaut MH. Handbook of Neurologic music therapy. Oxford: Oxford University Press; 2015.
- 37. Gerdner LA. Use of individualized music by trained staff and family: translating research into practice. J Gerontol Nurs 2005; 31(6): 22-30; quiz 55-6.
- 38.Gerdner LA. Effects of individualized versus classical "relaxation" music on the frequency of agitation in elderly persons with Alzheimer's disease and related disorders. Int Psychogeriatr 2000; 12(1): 49-65.
- 39. Theorell T. Psychological Health Effects of Musical Experiences. Theories, Studies and Reflections in Music Health Science. Heidelberg: Springerbriefs in Psychology; 2014.
- 40.Myskja A. Integrated music in nursing homes an approach to dementia care Bergen: University of Bergen; 2012.
- 41.Center for Disease Control and prevention. International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM).  $18.08.2017\ 2017$ . https://www.cdc.gov/nchs/icd/icd10cm.htm (accessed  $16.05\ 2018$ ).
- 42.Boell SK, Cecez-Kecmanovic D. Literature reviews and the hermeneutic circle. Australian Academic & Research Libraries 2010; 41(2): 129-44.
- 43. Craig P, Dieppe P, Macintyre S, et al. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ 2008; 337: a1655.
- 44. Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982; 140: 566-72.
- 45. Husebo BS, Strand LI, Moe-Nilssen R, Husebo SB, Snow AL, Ljunggren AE. Mobilization-Observation-Behavior-Intensity-Dementia Pain Scale (MOBID): development and validation of a nurse-administered pain assessment tool for use in dementia. J Pain Symptom Manage 2007; 34(1): 67-80.
- 46. Husebo BS, Strand LI, Moe-Nilssen R, Husebo SB, Ljunggren AE. Pain behaviour and pain intensity in older persons with severe dementia: reliability of the MOBID Pain Scale by video uptake. Scand J Caring Sci 2009; 23(1): 180-9.

- 47.Roen I, Selbaek G, Kirkevold O, Engedal K, Lerdal A, Bergh S. The Reliability and Validity of the Norwegian Version of the Quality of Life in Late-Stage Dementia Scale. Dement Geriatr Cogn Disord 2015; 40(3-4): 233-42.
- 48. Weiner MF, Martin-Cook K, Svetlik DA, Saine K, Foster B, Fontaine CS. The quality of life in late-stage dementia (QUALID) scale. J Am Med Dir Assoc 2000; 1(3): 114-6.
- 49.Brod M, Stewart AL, Sands L, Walton P. Conceptualization and measurement of quality of life in dementia: the dementia quality of life instrument (DQoL). Gerontologist 1999; 39(1): 25-35.
- 50. Barthel Activities of Daily Living (ADL) Index. Occas Pap R Coll Gen Pract 1993; (59): 24.
- 51. Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology1997;48: 10-6.
- 52.Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biological psychiatry 1988; 23(3): 271-84.
- 53. Husebo BS, Ballard C, Fritze F, Sandvik RK, Aarsland D. Efficacy of pain treatment on mood syndrome in patients with dementia: a randomized clinical trial. Int J Geriatr Psychiatry 2014; 29(8): 828-36.
- 54. Husebo BS, Ballard C, Sandvik R, Nilsen OB, Aarsland D. Efficacy of treating pain to reduce behavioural disturbances in residents of nursing homes with dementia: cluster randomised clinical trial. BMJ 2011; 343: d4065.
- 55.Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ  $2001;\ 323(7321):\ 1123-4.$